CLINICAL TRIAL: NCT06692010
Title: Comparison Between Clavipectoral Fascia Block & Interscalene Brachial Plexus Block As Regard Adequacy of Anesthesia in Clavicle Surgeries
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Sara Gamal Ibrahem Othman, Resident doctor at Anesthesia, Intensive Care and Pain Management department, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ISBP VS CPB Clavicle Surgeries
Record Dates: First submitted 2024-11-14; First posted 2024-11-18 (Actual); Last update posted 2024-11-18 (Actual); Status verified 2024-11

CONDITIONS: Clavicle Fracture
Keywords: Clavipectoral Fascia Block; Interscalene Brachial Plexus Block
MeSH Terms: interventions — Bupivacaine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Group CPB (Experimental): Clavipectoral fascia plane block group
  Interventions: Drug: Bupivacaine with Dexamethasone Solution
- Group ISBP & SCPB (Experimental): Interscalene brachial plexus block & superficial cervical plexus block group
  Interventions: Drug: Bupivacaine with Dexamethasone Solution

INTERVENTIONS:
Drug: Bupivacaine with Dexamethasone Solution — 10 to 15 ml %0.25 bupivacaine & 4 mg Dexamethazone

SUMMARY:
A newer technique called clavipectoral fascial plane block (CPB), introduced by Valdés-Vilches in 2017, involves injecting local anesthetic under ultrasound guidance between the clavipectoral fascia and periosteum at the injury site. This method offers a promising alternative for effective regional anesthesia in clavicular fracture surgeries. this study is aim to Comparison Between Use of Ultrasound guided Clavipectroal fascia block ( CPB ) & interscalene brachial plexus block ( ISBP ) As Regard Adeqacy of Anesthesia in clavicle Fracture

DETAILED DESCRIPTION:
Clavicle fractures represent 2.6% of all fractures and are commonly seen in emergency and surgical settings, particularly among young men due to sports or traffic incidents, predominantly affecting the mid-clavicle. Surgical intervention often yields better functional outcomes compared to conservative treatment. While general anesthesia is an option, it carries risks such as nausea, vomiting, and increased costs for patients. In contrast, regional anesthesia can effectively manage pain while minimizing complications associated with general anesthesia.

The supraclavicular nerve innervates the skin above the clavicle, but the sensory innervation of the clavicle itself remains debated. A combination of superficial cervical plexus block (SCPB) and interscalene brachial plexus block (ISBP) is frequently employed during clavicle fracture surgeries. The brachial plexus includes nerves from C5-8 and T1, while the cervical plexus comprises branches from both deep and superficial cervical structures. Although this combination can effectively address pain management during surgery, ISBP may lead to complications like diaphragmatic paralysis due to phrenic nerve involvement.

ELIGIBILITY:
Inclusion Criteria:

* . Patients who have isolated clavicle surgery. American Society of Anesthesiologists (ASA) classification I-II

Exclusion Criteria:

* 1.Patient with Major Trauma Insult " Brain \ chest \ Abdomen " 2.History of bleeding diathesis 3.Patients receiving anticoagulant treatment, 4.Patients known local anesthetics and opioid allergy, 5.Infection of the skin at the site of the needle puncture, 6.Pregnant or lactating females, 7.Patients who do not accept the procedure

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2024-12-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Pain Scores | 24 hours
  Postoperative pain level will be assessed using a visual analog scale (VAS) from (0 that's no pain to 10 that's unbearable pain) at specific time points (1, 6, 12, 24 hours post-surgery)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Fugelli CG, Westlye ET, Ersdal H, Strand K, Bjorshol C. Combined Interscalene Brachial Plexus and Superficial Cervical Plexus Nerve Block for Midshaft Clavicle Surgery: A Case Series. AANA J. 2019 Oct;87(5):374-378. PMID 31612842
- [Background] Atalay YO, Ciftci B, Ekinci M, Yesiltas S. The effectiveness of clavipectoral fascia plane block for analgesia after clavicle surgery: a report of five cases. Minerva Anestesiol. 2020 Sep;86(9):992-993. doi: 10.23736/S0375-9393.20.14503-6. Epub 2020 May 18. No abstract available. PMID 32420714